CLINICAL TRIAL: NCT06333093
Title: Optimization of Duodenal Tissue Resection Acquisition Study
Brief Title: Duodenal tIssue ResEction aCquisiTion (DIRECT) Study
Acronym: DIRECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jacques J.G.H.M. Bergman, Head of Endoscopy and Principle Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL82178.018.22
Record Dates: First submitted 2024-02-21; First posted 2024-03-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Duodenum Disease
MeSH Terms: conditions — Duodenal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cold snare resections (Experimental): Two (2) cold snare resections of the duodenal mucosa during an already scheduled upper gastrointestinal interventional endoscopy under deep sedation (propofol).
  Interventions: Procedure: Cold snare

INTERVENTIONS:
Procedure: Cold snare — Two (2) cold snare resections of the duodenal mucosa during an already scheduled upper gastrointestinal interventional endoscopy under deep sedation (propofol).

SUMMARY:
To evaluate the quality of cold snare resection specimens of duodenal mucosa tissue in patients undergoing an upper gastrointestinal interventional endoscopy in order to improve the processing of histological samples and its assessment in general and for future duodenal ablation studies.

DETAILED DESCRIPTION:
The duodenum plays an important role in metabolic health. There is evidence that the duodenal mucosa undergoes certain histological changes in the development of features of the metabolic syndrome and ultimately type 2 diabetes (T2D). To date, it is not known exactly what type of histological changes the duodenal mucosa undergoes in T2D, so elucidating these changes may lead to a better understanding and potentially new treatment options for metabolic syndrome and T2D.

The assessment of histological changes in tissue obtained from duodenal biopsies has proven to be very difficult due to the lack of orientation in the histological slides obtained. The investigators have learned that duodenal biopsies are too small and superficial to reliably assess histological changes in the duodenal mucosa and submucosa. Currently, the investigators are taking small cold snare resections from the duodenum to try to fully assess the duodenal (sub)mucosa. However, the investigators still have problems with the orientation of these resections. When slides are made, the specimens are curled, cut tangentially and artefacts occurr. As a result, it is still not possible to make a proper assessment of the duodenal (sub)mucosa.

Therefore, the investigators aim to optimise the process of obtaining, storing, processing and staining the duodenal mucosal tissue samples from cold snare resections. The investigators plan to optimise this process in patients who have already undergone upper gastrointestinal interventional endoscopy, including ablation therapy, endoscopic submucosal dissection (ESD) or endoscopic mucosal resection (EMR) for Barrett's neoplasia and squamous cell carcinoma of the oesophagus or small gastric neoplasia, or oesophageal dilatations, as the endoscopist performing DMR in the Netherlands also specialises in these endoscopic treatments. By studying the process of obtaining duodenal mucosal tissue samples in this specific patient population, there is no need to expose other patients to an upper gastrointestinal endoscopy with the associated propofol sedation.

ELIGIBILITY:
Inclusion Criteria:

* Already scheduled to undergo an upper gastrointestinal interventional endoscopy
* Endoscopy under deep sedation (propofol) in Amsterdam UMC

Exclusion Criteria:

* Previous GI surgery that could affect the ability to reach the duodenum via endoscopy, such as Bilroth 2, Roux-en-Y gastric bypass, or other similar procedures or condition
* History of duodenal inflammatory diseases including Crohn's Disease and Celiac Disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Acquiring larger pieces of tissue from the duodenum | 1 day
  Feasibility of acquiring adequate duodenual samples with the cold snare technique.
Histopatholocial assessment of larger pieces of tissue from the duodenum | 6 months
  Ability to histopathologically assess the tissue.
Checking if the tissue is of good quality enough for single cell RNA sequencing | 3 months
  The ability to dissociate the tissue to a sufficient degree to allow single cell RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques JG Bergman, MD PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Busch CBE, van den Hoek K, Neefjes-Borst EA, Nieuwdorp M, van Baar ACG, Bergman JJHGM. Optimizing duodenal tissue acquisition for mechanistic studies of duodenal ablation in type 2 diabetes. Endosc Int Open. 2025 Jan 29;13:a25032135. doi: 10.1055/a-2503-2135. eCollection 2025. PMID 40007651